CLINICAL TRIAL: NCT04049825
Title: A Phase 1, Multi-center, Open-label, Uncontrolled, Dose-escalation Trial to Evaluate the Safety of OPB-111077 in Combination With Bendamustine and Rituximab in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Phase 1 Trial of OPB-111077 in Combination With Bendamustine and Rituximab in Patients With r/r DLBCL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 317-102-00007; jRCT2080224718 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2019-07-09; First posted 2019-08-08 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Relapsed or Refractory Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Stage (Experimental): The dose of OPB-111077 in the first cohort will be 200 mg/day, increasing as appropriate to 400 mg/day in the second cohort and then to 600 mg/day in the third cohort.
  Interventions: Drug: OPB-111077
- Dose Expansion Stage (Experimental): 4 days on and 3days off of 21-day cycles of OPB-111077 Day 1 of 21-days cycles of rituximab Day 2 and 3 of 21-day cycles of bendamustine
  Interventions: Drug: OPB-111077

INTERVENTIONS:
Drug: OPB-111077 — OPB-111077+bendamustine
  Arms: Dose Escalation Stage
Drug: OPB-111077 — OPB-111077+rituximab+bendamustine
  Arms: Dose Expansion Stage

SUMMARY:
To investigate the tolerability and safety of OPB-111077 in combination with bendamustine and rituximab in patients with r/r DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definite diagnosis of Diffuse large B-cell lymphoma(DLBCL)
* Patients who have received at least initial standard treatment
* Patients with measurable lesions (based on International Working Group [IWG] 2014 criteria)
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1

<Only for dose-expansion stage>

* Patients who are pathologically diagnosed as CD20 positive lymphoma
* Patients who have a history of being treated with 1 to 5 regimens of previous chemotherapy for the underlying disease

Exclusion Criteria:

* Patients who are candidates for autologous or allogeneic hematopoietic stem cell transplantation
* Patients who were refractory to initial standard treatment
* Patients who have a history of bendamustine administration and are intolerant to bendamustine
* Patients with central nervous system (CNS) involvement of lymphoma or with a history of CNS involvement of lymphoma
* Patients diagnosed with DLBCL transformed from low-grade B-cell non-Hodgkin's lymphoma (NHL)

<Only for dose-expansion stage>

- Patients who have a history of rituximab administration and are intolerant to rituximab

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 23days
  The tolerability of OPB-111077 in combination with bendamustine and rituximab
Incidence of Adverse events(AEs) | Up to 3 years
  Safety of OPB-111077 in combination with bendamustine and rituximab

SECONDARY OUTCOMES:
Efficacy based on International working group(IWG) Lugano response criteria for Non Hodgkin's lymphoma ( (NHL) (2014)) | Last dose of study drug (up to 3 years)
  * Percentage of Participants with Complete Response based on International working group(IWG) Lugano response criteria for Non Hodgkin's lymphoma ( (NHL) (2014))
  * Percentage of Participants with Complete Response and Partial Response based on International working group(IWG) Lugano response criteria for Non Hodgkin's lymphoma ( (NHL) (2014))

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Yamagata University Hospital, Yamagata, Japan

IPD SHARING:
Plan to Share IPD: No
The focus of this study is a rare disease.